CLINICAL TRIAL: NCT01090804
Title: The Effectiveness of BreatheMAX Breathing Device on Airway Secretion Clearance in Patients With Ventilatory Dependence
Brief Title: The Effectiveness of BreatheMAX Breathing Device on Secretion Clearance
Acronym: ESMOSC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Khon Kaen university ( Graduate School ), Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 47660279
Record Dates: First submitted 2010-01-07; First posted 2010-03-23 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-01

CONDITIONS: Lung Disease
Keywords: BreatheMAX breathing device; Secretion clearance; Ventilatory dependence; Intubated patients
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- breathing exercise (Experimental): BreatheMAX breathing device is Water pressure Threshold Bottle. The level of water in the cylinder determines the load for treatment. In the treatment using 20% PNIP (Peak negative inspiratory pressure) was performed with 6-10 breaths/set; 10 set/day
  Interventions: Device: BreatheMAX breathing device

INTERVENTIONS:
Device: BreatheMAX breathing device — secretion clearance, breathing exercise

SUMMARY:
The purpose of this study is to determined effects of BreatheMAX on secretion clearance.

ELIGIBILITY:
Inclusion Criteria:

* One sign of secretion accumulation in bronchi
* Stable cardiopulmonary function
* Good consciousness and good co-operation

Exclusion Criteria:

* Massive hemoptysis
* Pneumothorax (untreated)

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
secretion wet weight (gram) | Three hours before, ten hours after treatment and night-time (02.00-07.00 am.)
  Airway mucus secretion was collected for three hours before and ten hours after treatment based on an auditory airway secretion sound and collected again at 02.00-07.00 am.The mucus secretion was collected by sterile suctioning technique via tracheostomy tube without adding any saline or sterile water.
viscosity of secretion | Three hours before and after treatment
  The secretion were collected in three hours before and after treatment, It were measured viscosity by First The mucus was gently homogenized by tissue grinder 5 ml (Cw11-205, Cowie, UK) for six minute at 37 degree celsius Second using Micro-Oswald viscometers with a capillary diameter of 0.77 mm for viscosity measure at same temperature in each sample(before and after).

SECONDARY OUTCOMES:
Heart rate (beat/min) | Before, during breathing exercise with device and immediate after treatment
  Heart rate was monitored before, during and immediate after breathing exercise with BreatheMAX (6-10 beats/set, 10 set/day and rest between ste for 1 minute)
Oxygen saturation (%SpO2) | Before, during breathing exercise with device and immediate after treatment
  Oxygen saturation was monitored before, during and immediate after breathing exercise with BreatheMAX (6-10 beats/set, 10 set/day and rest between set for 1 minute)
Respiratory rate (times/min) | In rest interval between set (1 minute)
  Respiratory rate was measured by manual for 1 minute before, rest interval between set and immediate after breathing exercise with device (during the patients reconnection mechanical ventilation)

CONTACTS AND LOCATIONS:
Overall Officials: Sujittra Kluayhomthong, Bachelor, Study Chair — Physical Therapy department, Faculty of Associated Medical Sciences, Khon Kaen university; Chulee CU Jones, Philosophy, Study Director — Physical Therapy Department, Faculty of Associated Medical Sciences, Khon Kaen university, Thailand; Wilaiwan Khrisanapant, Philosophy, Study Director — Department of physiology, Faculty of medicine, Khon Kaen university
Locations (1):
- Pulmonary research room of physical therapy department, Faculty of associated medical sciences, Khon Kaen University, Muang, Changwat Khon Kaen, Thailand